CLINICAL TRIAL: NCT07237074
Title: The Effect of Using Finger Puppets and Showing Cartoons on Pain and Fear in Preschool Children (3-6 Years Old) During Blood Collection
Brief Title: The Effect of Using Finger Puppets and Showing Cartoons on Pain and Fear in Preschool Children During Blood Collection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Zeynep Camkıran, nurse, Hitit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HititU-SBF-ZÇ-01
Record Dates: First submitted 2025-10-01; First posted 2025-11-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Fear; Pain
Keywords: blood collection; watching cartoons; finger puppet
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: three groups, including a cartoon and finger puppet group and a control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- finger puppet group (Experimental): During the blood collection procedure, 40 children were randomly selected to play with finger puppets.
  Interventions: Other: showing finger puppets during blood collection
- watching cartoons group (Experimental): During the blood collection procedure, 40 children were randomly selected to watch cartoons.
  Interventions: Other: cartoons
- control group (Experimental): No intervention was performed on the children.
  Interventions: Other: control group

INTERVENTIONS:
Other: showing finger puppets during blood collection — finger puppets
  Arms: finger puppet group
Other: cartoons — Watching cartoons during blood collection
  Arms: watching cartoons group
Other: control group — No intervention was made during blood collection
  Arms: control group

SUMMARY:
The study is a randomized controlled experimental study aimed at determining the effect of showing cartoons or using finger puppets to children aged 3-6 years before taking venous blood samples on their pain levels.

Based on the results of this study, it is thought that showing cartoons and using finger puppets before blood collection will help reduce pain levels in children and improve their ability to cope with pain, thereby improving the quality of care. In this context, the study will be conducted to determine the effect of showing cartoons and using finger puppets before blood collection on pain in pediatric patients.

DETAILED DESCRIPTION:
Children between the ages of three and six have the language skills to express pain at a sensory level. They can describe the location and intensity of the pain. They may cry, scream, and exhibit aggressive behavior in response to pain. They may think of invasive procedures such as blood collection as punishment. Before any procedures are performed, the child should be informed about the procedures that will be performed and their stress and fear should be reduced by helping them relax. Nurses should use non-pharmacological methods appropriate for the age group of the children during painful procedures to reduce the level of pain perceived by the children. In this study, I will examine the effect of showing cartoons and finger puppets to children during blood collection on pain and fear.

ELIGIBILITY:
Inclusion Criteria:

* The child and parent agree to participate in the study.
* The child is between 3 and 6 years old.
* The child has no acute pain complaints.
* The child has no disabilities.

Exclusion Criteria:

* The child and parent refuse to participate in the study.
* The child is under 3 years of age or over 6 years of age.
* The child has acute pain complaints.
* The child has any disability.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale | 4 months
  Pain scores are given according to the numerical values assigned to the faces on this scale. It is explained to the child that the faces on the scale do not represent people who are happy because they are not in pain or unhappy because they are in pain.
  A very happy person is Face 0. A little pain is Face 1, a little more pain is Face 2, a little more pain is Face 3, and quite a lot of pain is Face 4. Face 5 represents the highest level of pain that can be imagined. The child is asked to choose the face that best describes the pain they are feeling.
Children's Fear Scale (CFS) | 4 months
  CFS is used to score the fear that may cause pain in children before or during the procedure. The scale is a visual measurement tool consisting of five drawn lines ranging from a neutral facial expression (0 = no fear) to a frightened facial expression (4 = very afraid), with scores ranging from 0 to 4.
  The scale is used to assess the fear of pain in children before or during a procedure.
  The scale is a visual measurement tool consisting of five drawn lines ranging from a neutral facial expression (0 = no fear) to a frightened facial expression (4 = very afraid), with scores ranging from 0 to 4.
  The scale is used to assess the fear of pain in children before or during a procedure. . The Turkish language validity and psychometric properties of the scale used to assess procedural fears in children aged 5-12 were tested

SECONDARY OUTCOMES:
Information Form | 4 months
  Information Form: The form includes questions regarding the date of the procedure, the reason for the children's admission to the hospital, the duration of the procedure, the method used, the children's age, gender, whether they had received analgesics in the last 24 hours, whether they had undergone a blood draw in the last 6 months, whether any preparatory measures were taken before the blood draw and, if so, which method was used, the parents' age, family structure, and family education level.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Erol Olçok Education and Research Hospital, Çorum, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will not share the work data with anyone.